CLINICAL TRIAL: NCT01362933
Title: National Evaluation of the Adherence to Recommendations of VTE Treatment in Cancer Patients
Brief Title: National Evaluation of the Adherence to Recommendations of Venous Thrombo Embolism Treatment in Cancer Patients
Acronym: CARMEN
Status: Completed | Type: Observational
Sponsor: Floralis (Industry)
Collaborators: Centre Hospitalier Universitaire, Amiens (Other); Groupe Francophone Thrombose et Cancer (GFTC) (Unknown); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: Version N°2.0 du 21/03/2011
Record Dates: First submitted 2011-05-25; First posted 2011-06-01 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Neoplasms; Venous Thromboembolism
Keywords: PE; DVT; SVT; LMWH; VKA; international Venous Thromboembolism Recommendations
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VTE treatment in cancer patient: All patients with cancer present in the clinic, hospital, out patient diagnosed with a VTE during the 6 previous months.
  Interventions: Procedure: VTE treatment in cancer patient description

INTERVENTIONS:
Procedure: VTE treatment in cancer patient description — proportion of patients treated for evolutive VTE according to international recommendations

SUMMARY:
Treatment of venous thromboembolism in cancer patients is specific and has been validated in trials that favor the use of LMWH (Low Molecular Weight Heparin) instead of VKA (Vitamin K Antagonist) treatment during 6 months. International recommendations have diffused this option.It is necessary to evaluate the compliance of physicians to this treatment by measuring the number of patients with cancer treated with long term use of LMWH.

ELIGIBILITY:
Inclusion Criteria:

All patients with cancer present in the clinic, hospital, out patients diagnosed with a VTE during the 6 previous months. VTE can be symptomatic or asymptomatic, can be located close to a central line, and of any type (DVT, PE, SVT)

Exclusion Criteria:

* Patient already included in a trial studying antithrombotic therapy
* Patient refusing the study
* Patient under 18 and/or not competent to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with cancer present in the clinic, hospital, out patients diagnosed with a VTE during the 6 previous months
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the adherence to recommendations of VTE treatment in cancer patients | At baseline (J0)
  Proportion of patients treated for evolutive VTE according to international recommandations Patients could be hospitalised or could be out patient

SECONDARY OUTCOMES:
Evaluation of VTE disease according to cancer diagnosis (proportion of SVT (Superficial Venous Thrombosis), DVT (Deep Venous Thrombosis), PE (Pulmonary Embolism) | At baseline (J0)
  Percentage of VTE (PE,DVT,SVT)and cancer type
Proportion of asymptomatic VTE disease for this population | At baseline (J0)
  percentage of VTE and cancer status (local, metastatic)
Feasibility of self injections for VTE treatment in cancer patients. | At baseline (J0)
  percentage of patients practising self injections
Proportion of patients with catheter thrombosis | At baseline (J0)
  Percentage of patients receiving novel cancer therapies

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Antoinette SEVESTRE, MD, Principal Investigator — Centre Hospitalier Universitaire, Amiens; Dominique FARGE BANCEL, MD, Study Director — GFTC; Jean Luc BOSSON, MD, Study Director — University Hospital, Grenoble
Locations (49):
- France (49):
  - CHR Annecy, Annecy
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CH AUCH, Auch
  - CH Beauvais, Beauvais
  - Institut Bergonie, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - Centre François Baclesse, Caen
  - CH Antoine Gayraud Cedex 9, Carcassonne
  - Clinique du Parc CASTELNAU LE LEZ, Castelnau-le-Lez
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - CH Chalons En Champagne, Châlons-en-Champagne
  - Centre Jean Perrin Clcc, Clermont-Ferrand
  - CHU, Clermont-Ferrand
  - Hopital Louis Mourier Colombes, Colombes
  - Polyclinique Saint come, Compiègne
  - CHU Bocage Dijon, Dijon
  - CHU, Grenoble
  - Ch Versailles Andre Maginot, Le Chesnay
  - CHRU Calmette, Lille
  - CHRU LILLE, Hôpital Huriez, Lille
  - CHRU Albert Calmette, Lille
  - Centre Hospitalier Edouard Herriot, Lyon
  - Hopital Desgenettes LYON, Lyon
  - Centre Leon Berard LYON, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Institut Paoli Calmette Marseille, Marseille
  - Hopital Saint Joseph, Marseille
  - CHU La Timone Marseille, Marseille
  - Hôpital Nord Marseille, Marseille
  - Centre Régional de Lutte Contre le Cancer Val d'Aurelle, Montpellier
  - CHU Hôtel-Dieu NANTES, Nantes
  - Centre de Lutte contre le Cancer (Centre René Gauducheau), Nantes
  - CHR Orleans, Orléans
  - Hopital Saint Louis Paris, Paris
  - Hopital Saint Antoine Paris, Paris
  - Hopital de la Salpetriere Paris, Paris
  - Hopital Val de GRACE, Paris
  - Hôpital Kremlin Bicêtre, Paris
  - CH Lyon Sud, Pierre-Bénite
  - CHU Rouen, Rouen
  - Centre Rene Hugunin institut curie, Saint-Cloud
  - Centre Hospitalier Mutualiste Site Etienne Dolet, Saint-Nazaire
  - Clinique Charcot,, Sainte-Foy-lès-Lyon
  - CHRU Strasbourg, Strasbourg
  - CH Valence, Valence
  - Ch Bretagne Atlantique, Vannes
  - Centre Hospitalier de Villefranche sur Saône, Villefranche-sur-Saône
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Frequency, risk factors, and trends for venous thromboembolism among hospitalized cancer patients. Cancer. 2007 Nov 15;110(10):2339-46. doi: 10.1002/cncr.23062. PMID 17918266
- [Background] Levitan N, Dowlati A, Remick SC, Tahsildar HI, Sivinski LD, Beyth R, Rimm AA. Rates of initial and recurrent thromboembolic disease among patients with malignancy versus those without malignancy. Risk analysis using Medicare claims data. Medicine (Baltimore). 1999 Sep;78(5):285-91. doi: 10.1097/00005792-199909000-00001. PMID 10499070
- [Background] Khorana AA, Francis CW, Culakova E, Lyman GH. Risk factors for chemotherapy-associated venous thromboembolism in a prospective observational study. Cancer. 2005 Dec 15;104(12):2822-9. doi: 10.1002/cncr.21496. PMID 16284987
- [Background] Blom JW, Vanderschoot JP, Oostindier MJ, Osanto S, van der Meer FJ, Rosendaal FR. Incidence of venous thrombosis in a large cohort of 66,329 cancer patients: results of a record linkage study. J Thromb Haemost. 2006 Mar;4(3):529-35. doi: 10.1111/j.1538-7836.2006.01804.x. PMID 16460435
- [Background] Chew HK, Wun T, Harvey D, Zhou H, White RH. Incidence of venous thromboembolism and its effect on survival among patients with common cancers. Arch Intern Med. 2006 Feb 27;166(4):458-64. doi: 10.1001/archinte.166.4.458. PMID 16505267
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Lee AY, Levine MN, Butler G, Webb C, Costantini L, Gu C, Julian JA. Incidence, risk factors, and outcomes of catheter-related thrombosis in adult patients with cancer. J Clin Oncol. 2006 Mar 20;24(9):1404-8. doi: 10.1200/JCO.2005.03.5600. PMID 16549834
- See also: American Society of Clinical Oncology guideline: recommendations for venous thromboembolism prophylaxis and treatment in patients with cancer. — http://www.ncbi.nlm.nih.gov/pubmed/17968019